CLINICAL TRIAL: NCT04929249
Title: A Randomized, Multicenter, Open-label Trial Comparing the Effectiveness of an "Inclisiran First" Implementation Strategy to Usual Care on LDL Cholesterol (LDL-C) in Patients With Atherosclerotic Cardiovascular Disease and Elevated LDL-C (≥70 mg/dL) Despite Receiving Maximally Tolerated Statin Therapy (VICTORION-INITIATE)
Brief Title: A Randomized Study to Evaluate the Effect of an "Inclisiran First" Implementation Strategy Compared to Usual Care in Patients With Atherosclerotic Cardiovascular Disease and Elevated LDL-C Despite Receiving Maximally Tolerated Statin Therapy (VICTORION-INITIATE)
Acronym: V-INITIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839A1US02
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Hyperlipidemia; Secondary Cardiovascular Prevention; Atherosclerotic Cardiovascular Disease (ASCVD); Hypercholesterolemia; Lipid lowering therapies; Inclisiran
MeSH Terms: conditions — Atherosclerosis; Hyperlipidemias; Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: randomized, two-arm, parallel-group, open-label, multicenter clinical trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran First (Experimental): Inclisiran sodium 300 mg 1.5 ml (equivalent to 284 mg of inclisiran) + usual care
  Interventions: Drug: Inclisiran
- Usual Care (No Intervention): Treating physicians were recommended to treat patients in accordance with the 2018 ACC/AHA guidelines

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300 mg/1.5 ml (equivalent to 284 mg inclisiran liquid) in prefilled syringe (PFS).
  Other Names: Inclisiran First
  Arms: Inclisiran First

SUMMARY:
The purpose of this study was to assess the effectiveness of an "inclisiran first" implementation strategy (addition of inclisiran to maximally tolerated statin therapy immediately upon failure to achieve acceptable LDL-C with maximally tolerated statin therapy alone) compared to usual care in an atherosclerotic cardiovascular disease (ASCVD) population.

DETAILED DESCRIPTION:
The study design was a randomized, two-arm, parallel-group, open-label, multicenter, clinical trial comparing an "inclisiran first" implementation strategy to usual care (1:1 randomization) with established ASCVD and elevated LDL-C (or non-HDL-C) despite treatment with maximally tolerated statin therapy.

Eligible patients had established ASCVD and elevated LDL-C levels ≥ 70 mg/dL (or non-HDL-C ≥ 100 mg/dL) despite treatment with maximally tolerated statin therapy.

In the "inclisiran first" implementation strategy group post-randomization, addition of other non-statin LDL-C lowering therapies (e.g., ezetimibe or bempedoic acid, excluding PCSK9 inhibiting monoclonal antibodies) were allowed to reach acceptable LDL-C levels. In the "inclisiran first" implementation strategy group, inclisiran was administered initially at randomization, 90 days later, and six months, thereafter.

ELIGIBILITY:
Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Males and females ≥18 years of age
3. History of ASCVD, documented by hospital records, claims data and/or prior laboratory/imaging assessments a Coronary heart disease (CHD):

   * Prior myocardial infarction
   * Prior coronary revascularization (PCI or CABG)
   * Angiographic or CT-imaging (e.g., MDCT/CTA) evidence of coronary atherosclerosis (>70% stenosis in at least one major epicardial coronary artery) b Cerebrovascular disease:
   * Prior ischemic stroke confirmed by a brain imaging study, CT or MRI; thought not to be caused by atrial fibrillation, valvular heart disease or mural thrombus
   * Carotid artery stenosis >70% on prior angiography or ultrasound
   * History of prior percutaneous or surgical carotid artery revascularization c Peripheral arterial disease (PAD):
   * Prior documentation of a resting ankle-brachial index ≤0.85
   * History of prior percutaneous or surgical revascularization of an iliac, femoral, or popliteal artery or aortic aneurysm
   * Prior non-traumatic amputation of a lower extremity due to peripheral artery disease
4. Serum LDL-C ≥70 mg/dL or non-HDL-C ≥100 mg/dL
5. Fasting triglyceride <5.65 mmol/L (<500 mg/dL) at screening
6. Calculated glomerular filtration rate >30 mL/min by estimated glomerular filtration rate (eGFR) using standardized local clinical methodology
7. Participants should be on maximally tolerated statin therapy, as determined by the investigator, with no immediate plans to modify lipid lowering therapies. Statin intolerant patients are eligible if they had documented side effects on at least 2 different statins, including one at the lowest standard dose
8. Participants must be willing and able to give informed consent before initiation of any study related procedures and willing to comply with all required study procedures

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study.

1. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the participant at significant risk (according to investigator's [or delegate] judgment) if he/she participates in the clinical study
2. An underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate) might interfere with interpretation of the clinical study results
3. New York Heart Association (NYHA) class III or IV heart failure or last known left ventricular ejection fraction <30%
4. Significant cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication or via ablation at the time of screening
5. Major adverse cardiovascular event within 6 months prior to randomization
6. Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization despite antihypertensive therapy
7. Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 2 years
8. History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the two years prior to randomization
9. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of investigational drug. Basic contraception methods include:

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
   3. Male sterilization (at least 6 m prior to screening). For female participants in the study, the vasectomized male partner should be the sole partner for that participant
   4. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps)
   5. Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.

   Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
10. Known history of alcohol and/or drug abuse within the last 5 years (occasional casual users of illicit drugs in the opinion of the investigators are not excluded)
11. Treatment with other investigational products or devices within 30 days or five half-lives of the screening visit, whichever is longer
12. History of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes
13. Planned use of other investigational products or devices during the course of the study
14. Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:

    1. Participants who are unable to communicate or to cooperate with the investigator
    2. Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including participants whose cooperation is doubtful due to drug abuse or alcohol dependency)
    3. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study - including potential participants who indicate that their participation is contingent on receiving inclisiran)
    4. Have any medical or surgical condition, which in the opinion of the investigator would put the participant at increased risk from participating in the study
    5. Persons directly involved in the conduct of the study
15. Previous or current treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9 or ezetimibe
16. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or alanine aminotransferase (ALT) elevation >3x ULN, aspartate aminotransferase (AST) elevation >3x ULN, or total bilirubin elevation >2x ULN (except patients with Gilbert's syndrome) at screening confirmed by a repeat measurement at least one week apart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (43):
  - ARcare Center for Clinical Research ., Little Rock, Arkansas
  - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Keck Medical Center USC ., Los Angeles, California
  - d-b-a Greenwich Cardio Assoc CLCZ696BUS08, Greenwich, Connecticut
  - Cardiology Ass of Fairfield County ., Stamford, Connecticut
  - Integrative Research Associates Inc, Fort Lauderdale, Florida
  - Elite Cardiac Research Center ., Hialeah, Florida
  - University of Florida Health Science Center ., Jacksonville, Florida
  - Jacksonville Ctr for Clin Rea Encore Research Group, Jacksonville, Florida
  - Internal Medicine and Cardiology, Kissimmee, Florida
  - Gateway Cardiology PC CACZ885M2301_Younis, Jerseyville, Illinois
  - Affinity Health Corp, Oak Brook, Illinois
  - Northwestern Medicine Northwestern University ., Winfield, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - St Elizabeth Healthcare ., Edgewood, Kentucky
  - Alexandria Cardiology Clinic ., Alexandria, Louisiana
  - Medstar Health Research Institute ., Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Bryan LGH Heart Inst Intigrated Cardiology Group ., Lincoln, Nebraska
  - Inspira Health Network The Heart House, Elmer, New Jersey
  - New Jersey Heart, Linden, New Jersey
  - New York Presbyterian Queens ., Flushing, New York
  - New York Presbyterian Hospital ., New York, New York
  - State Uni of NY at Stony Brook ., Stony Brook, New York
  - Montefiore Hospital ., The Bronx, New York
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Capital Area Research LLC Suite 330, Newport, Pennsylvania
  - Capital Area Research, Newport, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Alliance for Multispecialty Res LLC, Nashville, Tennessee
  - Cypress Heart and Vascular Center, Cypress, Texas
  - NW Houston Neuro Comp Sleep Med Ctr, Cypress, Texas
  - Primecare Medical Group, Houston, Texas
  - Synergy Group Medical LLC ., Houston, Texas
  - Synergy Group Medical LLC, Houston, Texas
  - Northwest Houston Cardiology PA ., Houston, Texas
  - Synergy Groups Medical LLC, Missouri City, Texas
  - Bay Area Heart Ace Clinical Resh Gp ., Webster, Texas
  - Centra Health ., Lynchburg, Virginia
  - National Clinical Research ., Richmond, Virginia
  - Exemplar Research Inc ., Morgantown, West Virginia
  - Marshfield Medical Clinic ., Marshfield, Wisconsin
  - Marshfield Clinic Health System, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Koren MJ, Rodriguez F, East C, Toth PP, Watwe V, Abbas CA, Sarwat S, Kleeman K, Kumar B, Ali Y, Jaffrani N. An "Inclisiran First" Strategy vs Usual Care in Patients With Atherosclerotic Cardiovascular Disease. J Am Coll Cardiol. 2024 May 21;83(20):1939-1952. doi: 10.1016/j.jacc.2024.03.382. Epub 2024 Apr 7. PMID 38593947
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 43 centers in the United States
Period: Overall Study
Arm/Group | Inclisiran First | Usual Care
Started | 225 | 225
Full Analysis Set (FAS) (The Full Analysis Set (FAS) comprised of all randomized patients. According to the intent to treat principle, patients were analyzed according to the treatment group they were assigned to during the randomization period.) | 225 | 225
Safety Set (The Safety Set included all patients who received study treatment. Patients were analyzed according to the study treatment received. Patients in the usual care treatment group who had data collected at the Baseline Visit were included in the safety set.) | 234 (Patients who were randomized to usual care and still received inclisiran as a concomitant medication any time during the course of the study were analyzed as part of the inclisiran first group.) | 216 (Including participants randomized to inclisiran first who did not receive inclisiran)
Completed | 212 | 195
Not Completed | 13 | 30
Not completed — Adverse Event | 2 | 1
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 3 | 11
Not completed — Technical problems | 0 | 1
Not completed — Subject decision | 6 | 8
Not completed — Withdrew consent | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran First | Usual Care | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.01) | 66.8 (9.84) | 66.5 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 139
  Male | 158 | 153 | 311
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 186 | 187 | 373
  Black or African American | 27 | 29 | 56
  Asian | 8 | 4 | 12
  Unknown | 4 | 4 | 8
  Multiple | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C
Description: Percent change from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) of an "inclisiran first" implementation strategy compared to usual care at Day 330.
Time Frame: Baseline, Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients. Number of participants analyzed corresponds to the number of subjects who had LDL-C values at baseline and Day 330.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: percent change in LDL-C
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 205 | 174
percent change in LDL-C | -60.0 [-64.7 to -55.2] | -7.0 [-12.0 to -1.9]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -53.0, 97.5% CI 2-sided [-60.0 to -46.0]

2. Primary Outcome: Percentage of Participants Who Discontinued Statin Therapy
Description: Percentage of patients who discontinued statin therapy ≥ 30 days before the end-of-study visit of an "inclisiran first" implementation strategy compared to usual care, for patients in the FAS excluding those with a medical history of statin intolerance.
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients. Participants with Medical History of Statin Intolerance were excluded from this analysis.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 166 | 168
Percentage of participants | 6.0 [1.9 to 10.2] | 16.7 [10.2 to 23.1]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Non-Inferiority — Non-inferiority was declared if the upper limit of the one-sided 98.75% confidence interval did not exceed the non-inferiority margin of 15%; Normal approx. to binomial distribution; Difference in percentage = -10.6, 97.5% CI 2-sided [-18.3 to -3.0]; Upper limit of one-sided 98.75% CI (-3.0%)

3. Secondary Outcome: Absolute Change From Baseline in LDL-C
Description: Absolute change in Low-Density Lipoprotein Cholesterol (LDL-C) of an "inclisiran first" implementation strategy compared to usual care at Day 330
Time Frame: Baseline, Day 330
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 205 | 174
mg/dL | -58.0 [-61.6 to -54.4] | -10.5 [-14.3 to -6.6]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -47.6, 95% CI 2-sided [-52.8 to -42.3]

4. Secondary Outcome: Average Percent Change From Baseline in LDL-C Levels Across Visits
Description: Average percent change in Low-Density Lipoprotein Cholesterol (LDL-C) of an "inclisiran first" implementation strategy compared to usual care across visits.
  Calculated by averaging the observed post-baseline values (percent change) for each participant across analysis visits.
Time Frame: Up to 330 Days
Population: Full Analysis Set (FAS) comprised of all randomized patients. Number of participants analyzed corresponds to the number of subjects who had LDL-C average change from baseline values.
Measure: Least Squares Mean (95% Confidence Interval); unit: Average percent change in LDL-C
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 222 | 209
Average percent change in LDL-C | -57.2 [-60.3 to -54.0] | -2.8 [-6.0 to 0.5]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Linear; LS mean difference = -54.4, 95% CI 2-sided [-59.0 to -49.8]

5. Secondary Outcome: Average Absolute Change From Baseline in LDL-C Levels Across Visits
Description: Average absolute change in Low-Density Lipoprotein Cholesterol (LDL-C) of an "inclisiran first" implementation strategy compared to usual care across visits.
  Calculated by averaging the observed post-baseline values (absolute change) for each participant across analysis visits.
Time Frame: Up to 330 days
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 222 | 209
mg/dL | -55.0 [-57.8 to -52.2] | -6.0 [-8.9 to -3.2]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Linear; LS mean difference = -48.9, 95% CI 2-sided [-52.9 to -44.9]

6. Secondary Outcome: Percentage of Participants Achieving ≥ 50% Reduction From Baseline in LDL-C
Description: Percentage of patients achieving a ≥ 50% reduction from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) levels of an "inclisiran first" implementation strategy compared to usual care at Day 330.
  Missing data is imputed using "non-responder" (i.e., "negative" outcome) imputation.
Time Frame: Baseline, Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 225 | 225
Percentage of participants | 69.8 | 5.3
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 42.32, 95% CI 2-sided [22.07 to 81.16]

7. Secondary Outcome: Percentage of Participants Achieving LDL-C < 100 mg/dL.
Description: Percentage of participants achieving Low-Density Lipoprotein Cholesterol (LDL-C) < 100 mg/dL (among the subset of participants with LDL-C >=100 mg/dL at baseline) of an "inclisiran first" implementation strategy compared to usual care at Day 330.
  Missing data is imputed using "non-responder" (i.e., "negative" outcome) imputation.
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients. Only a subset of participants with LDL-C >=100 mg/dL at baseline were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 77 | 81
Percentage of participants | 80.5 | 32.1
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.32, 95% CI 2-sided [6.72 to 44.66]

8. Secondary Outcome: Percentage of Participants Achieving LDL-C < 70 mg/dL
Description: Percentage of participants achieving Low-Density Lipoprotein Cholesterol (LDL-C) < 70 mg/dL of an "inclisiran first" implementation strategy compared to usual care at Day 330.
  Missing data is imputed using "non-responder" (i.e., "negative" outcome) imputation.
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 225 | 225
Percentage of participants | 81.8 | 22.2
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 24.46, 95% CI 2-sided [14.18 to 42.19]

9. Secondary Outcome: Percentage of Participants Achieving LDL-C < 55 mg/dL
Description: Percentage of participants achieving Low-Density Lipoprotein Cholesterol (LDL-C) < 55 mg/dL of an "inclisiran first" implementation strategy compared to usual care at Day 330.
  Missing data is imputed using "non-responder" (i.e., "negative" outcome) imputation.
Time Frame: Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 225 | 225
Percentage of participants | 71.6 | 8.9
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 35.12, 95% CI 2-sided [19.51 to 63.24]

10. Secondary Outcome: Percent Change in Lipids and Other Lipoproteins From Baseline
Description: Percent change in plasma lipids, lipoproteins and triglycerides in participants receiving an "inclisiran first" implementation strategy compared to usual care at Day 330
Time Frame: Baseline, Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients. Number of participants analyzed corresponds to the number of subjects who had values at baseline and Day 330.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 208 | 178
Percent change
  Total Cholesterol | -34.1 [-36.7 to -31.6] | -4.1 [-6.8 to -1.4]
  HDL Cholesterol: number analyzed (Participants) | 208 | 177
  HDL Cholesterol | 8.5 [6.5 to 10.6] | 2.0 [-0.2 to 4.2]
  Non-HDL Cholesterol: number analyzed (Participants) | 207 | 177
  Non-HDL Cholesterol | -49.3 [-52.7 to -46.0] | -5.1 [-8.7 to -1.6]
  VLDL Cholesterol: number analyzed (Participants) | 207 | 176
  VLDL Cholesterol | -10.1 [-14.8 to -5.4] | 6.8 [1.8 to 11.9]
  Triglycerides: number analyzed (Participants) | 208 | 177
  Triglycerides | -10.6 [-15.3 to -5.9] | 7.2 [2.1 to 12.2]
  Apolipoprotein B: number analyzed (Participants) | 203 | 176
  Apolipoprotein B | -46.4 [-49.7 to -43.1] | -3.8 [-7.3 to -0.3]
  Lipoprotein(a): number analyzed (Participants) | 201 | 178
  Lipoprotein(a) | -19.6 [-22.2 to -16.9] | 2.3 [-0.5 to 5.2]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Total Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -30.1, 95% CI 2-sided [-33.8 to -26.3]
Statistical Analysis 2: Comparison: Inclisiran First vs Usual Care; HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = 6.6, 95% CI 2-sided [3.6 to 9.5]
Statistical Analysis 3: Comparison: Inclisiran First vs Usual Care; Non-HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -44.2, 95% CI 2-sided [-49.1 to -39.3]
Statistical Analysis 4: Comparison: Inclisiran First vs Usual Care; VLDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -16.9, 95% CI 2-sided [-23.8 to -10.0]
Statistical Analysis 5: Comparison: Inclisiran First vs Usual Care; Triglycerides; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -17.8, 95% CI 2-sided [-24.7 to -10.9]
Statistical Analysis 6: Comparison: Inclisiran First vs Usual Care; Apolipoprotein B; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -42.6, 95% CI 2-sided [-47.5 to -37.8]
Statistical Analysis 7: Comparison: Inclisiran First vs Usual Care; Lipoprotein(a); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -21.9, 95% CI 2-sided [-25.8 to -18.0]

11. Secondary Outcome: Absolute Change in Lipids and Other Lipoproteins From Baseline
Description: Absolute change in plasma lipids, lipoproteins and triglycerides in participants receiving an "inclisiran first" implementation strategy compared to usual care at Day 330
Time Frame: Baseline, Day 330
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 208 | 178
mg/dL
  Total Cholesterol | -59.6 [-63.8 to -55.5] | -9.7 [-14.1 to -5.2]
  HDL Cholesterol: number analyzed (Participants) | 208 | 177
  HDL Cholesterol | 3.5 [2.6 to 4.4] | 0.3 [-0.6 to 1.3]
  Non-HDL Cholesterol: number analyzed (Participants) | 207 | 177
  Non-HDL Cholesterol | -63.0 [-66.9 to -59.1] | -10.5 [-14.7 to -6.4]
  VLDL Cholesterol: number analyzed (Participants) | 207 | 176
  VLDL Cholesterol | -4.6 [-5.9 to -3.4] | 0.0 [-1.4 to 1.3]
  Triglycerides: number analyzed (Participants) | 208 | 177
  Triglycerides | -25.4 [-31.9 to -18.9] | -0.1 [-7.0 to 6.8]
  Apolipoprotein B: number analyzed (Participants) | 203 | 176
  Apolipoprotein B | -43.6 [-45.9 to -41.3] | -7.3 [-9.8 to -4.8]
  Lipoprotein(a): number analyzed (Participants) | 201 | 178
  Lipoprotein(a) | -9.8 [-11.1 to -8.4] | -1.0 [-2.5 to 0.4]
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Total Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -49.9, 95% CI 2-sided [-56.0 to -43.9]
Statistical Analysis 2: Comparison: Inclisiran First vs Usual Care; HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = 3.1, 95% CI 2-sided [1.8 to 4.4]
Statistical Analysis 3: Comparison: Inclisiran First vs Usual Care; Non-HDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -52.4, 95% CI 2-sided [-58.1 to -46.7]
Statistical Analysis 4: Comparison: Inclisiran First vs Usual Care; VLDL Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -4.6, 95% CI 2-sided [-6.5 to -2.8]
Statistical Analysis 5: Comparison: Inclisiran First vs Usual Care; Triglycerides; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -25.3, 95% CI 2-sided [-34.8 to -15.8]
Statistical Analysis 6: Comparison: Inclisiran First vs Usual Care; Apolipoprotein B; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -36.3, 95% CI 2-sided [-39.7 to -32.9]
Statistical Analysis 7: Comparison: Inclisiran First vs Usual Care; Lipoprotein(a); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS mean difference = -8.7, 95% CI 2-sided [-10.7 to -6.8]

12. Secondary Outcome: Percentage of Participants by Intensity of Lipid Lowering Therapy
Description: Percentage of participants with decrease in dose, no change in dose or increase in dose to assess changes in background lipid-lowering therapy in participants receiving an "inclisiran first" implementation strategy compared to usual care at Day 330
Time Frame: Baseline, Day 330
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 215 | 199
Percentage of participants
  Decrease in statin intensity | 2.3 | 4.5
  No change in statin intensity | 97.2 | 93.0
  Increase in statin intensity | 0.5 | 2.5
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p = 0.899, proportional odds model; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.43 to 2.61]

13. Secondary Outcome: Proportion of Days Covered by Medication
Description: Proportion of days covered refers to the total number of days on either statin, ezetimibe, bempedoic acid or PCSK9 inhibiting monoclonal antibody therapies taken during the study divided by total number of study days, calculated for each participant; If a participant did not take any of the four medications then the total number of days will be assumed to be zero.
Time Frame: Up to 330 Days
Population: Full Analysis Set (FAS) comprised of all randomized patients. Participants with missing baseline LDL-C are excluded from the regression analysis.
Measure: Least Squares Mean (Standard Error); unit: proportion of days covered
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 224 | 224
proportion of days covered | 0.894 (0.0169) | 0.902 (0.0169)
Statistical Analysis 1: Comparison: Inclisiran First vs Usual Care; Test type: Superiority; p = 0.727, Regression, Linear; LS mean difference = -0.008, 95% CI 2-sided [-0.055 to 0.039]

14. Secondary Outcome: LDL-C Measures of Variability - Standard Deviation
Description: Visit-to-visit LDL-C variability from Day 90 until Day 330 of an "inclisiran first" implementation strategy compared to usual care. It was assessed using two measures of variability: standard deviation and coefficient of variation.
Time Frame: Day 90, Day 180, Day 270 and Day 330
Population: Full Analysis Set (FAS) comprised of all randomized patients. Number of participants analyzed corresponds to the number of subjects who had available values at each timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 213 | 201
mg/dL
  Day 90 | 42.6 (27.21) | 94.3 (38.33)
  Day 180: number analyzed (Participants) | 207 | 191
  Day 180 | 41.1 (28.39) | 91.2 (31.61)
  Day 270: number analyzed (Participants) | 204 | 178
  Day 270 | 46.2 (31.22) | 88.4 (32.16)
  Day 330: number analyzed (Participants) | 205 | 174
  Day 330 | 38.8 (25.33) | 86.8 (35.47)

15. Secondary Outcome: LDL-C Measures of Variability - Coefficient of Variation
Description: as for outcome 14
Time Frame: Day 90, Day 180, Day 270 and Day 330
Population: as for outcome 14
Measure: Number; unit: Coefficient of Variation
Arm/Group | Inclisiran First | Usual Care
Number analyzed (Participants) | 213 | 201
Coefficient of Variation
  Day 90 | 63.90 | 40.65
  Day 180: number analyzed (Participants) | 207 | 191
  Day 180 | 69.00 | 34.67
  Day 270: number analyzed (Participants) | 204 | 178
  Day 270 | 67.56 | 36.38
  Day 330: number analyzed (Participants) | 205 | 174
  Day 330 | 65.34 | 40.89

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 330 days or until resolution.
Description: All safety analyses were conducted in the Safety Set.
Arm/Group | Inclisiran First | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/234 | 1/216
Serious Adverse Events (participants affected / at risk) | 27/234 | 29/216
Other Adverse Events (participants affected / at risk) | 64/234 | 53/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran First (N=234) | Usual Care (N=216)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Viral pericarditis (Infections and infestations) | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood parathyroid hormone increased (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal ganglia stroke (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 2 | 1
Middle cerebral artery stroke (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal atrophy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran First (N=234) | Usual Care (N=216)
Injection site pain (General disorders) | 18 | 0
COVID-19 (Infections and infestations) | 18 | 14
Urinary tract infection (Infections and infestations) | 8 | 7
Fall (Injury, poisoning and procedural complications) | 3 | 9
Blood creatine phosphokinase increased (Investigations) | 10 | 13
Glycosylated haemoglobin increased (Investigations) | 9 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04929249/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT04929249/SAP_001.pdf